CLINICAL TRIAL: NCT05253820
Title: Comparison of the Long-term Radial Artery Occlusion in Coronary Diagnosis and Intervention Via Distal vs Conventional Radial Approach: Randomized-controlled Trial(CONDITION)
Brief Title: Long-term Radial Artery Occlusion in Coronary Diagnosis and Intervention Via Distal Radial Approach (CONDITION)
Acronym: CONDITION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wujin People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20220130
Record Dates: First submitted 2022-02-03; First posted 2022-02-24 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Coronary Artery Disease; Distal Radial Artery; Radial Artery Occlusion
Keywords: coronary artery disease; distal radial artery; conventional radial artery; radial artery occlusion
MeSH Terms: conditions — Coronary Artery Disease; Arterial Occlusive Diseases

STUDY DESIGN:
Intervention Model Description: Single-center parallel randomized controlled study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- distal radial approach group (Experimental): subjects randomized to experimental group were underwent coronary diagnosis and intervention via distal radial approach
  Interventions: Procedure: distal radial approach
- conventional radial access group (Active Comparator): subjects randomized to active comparator group were underwent coronary diagnosis and intervention via conventional radial approach
  Interventions: Procedure: conventional radial access

INTERVENTIONS:
Procedure: distal radial approach — coronary diagnosis and intervention via distal vs conventional radial approach
  Arms: distal radial approach group
Procedure: conventional radial access — conventional radial access
  Arms: conventional radial access group

SUMMARY:
Randomized-controlled trial to comparison of the long-term radial artery occlusion in coronary diagnosis and intervention via distal vs conventional radial approach

DETAILED DESCRIPTION:
Coronary diagnosis and intervention via distal radial artery is prevalent worldwide. This study aims to explore the long-term radial artery occlusion after coronary diagnosis and intervention via distal radial artery at 3 months after procedure using portable high-frequent ultrasound. The secondary endpoints include the success rate of puncture, time of puncture, duration of hemostasis, radial artery trauma, etc.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Palpable unilateral distal radial and radial artery

Exclusion Criteria:

* Age ≥ 90years;
* Height≥ 185cm;
* Cardiogenic shock;
* Contraindications to puncture at the puncture site;
* Inability to obtain written informed consent
* Previous right radial or distal artery intervention

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 801 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
long-term radial artery occlusion | 3 months after procedure
  Number of participants with the forearm radial artery occlusion is detected using high-frequent ultrasound at 3 months after procedure

SECONDARY OUTCOMES:
radial artery occlusion | at 24 hours after procedure
  Number of participants with the forearm radial artery occlusion is detected using high-frequent ultrasound at 24 hours after procedure
success rate of puncture | at 24 hours post procedure
  Success of puncture is defined as the sheath inserted into the artery
time of puncture | at 24 hours post procedure
  time of puncture is defined as the time from initial puncture to the sheath inserted into the artery
Radial artery trauma | at 24 hours and 3 months post procedure
  Number of participants with radial artery trauma in the radial and distal radial artery, such as the intimal tears, dissections, thrombosis, and pseudoaneurysms in the radial and distal radial artery, which is detected by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Gaojun Cai, MD, Study Chair — Cardiovascular department, Changzhou Wujin People's Hospital
Locations (1):
- Changzhou Wujin People's Hospital, Changzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gupta A, Agstam S. Radial Artery Pseudoaneurysm Following Percutaneous Coronary Intervention. J Invasive Cardiol. 2021 May;33(5):E406. doi: 10.25270/jic/20.00272. PMID 33932290
- [Result] Rashid M, Kwok CS, Pancholy S, Chugh S, Kedev SA, Bernat I, Ratib K, Large A, Fraser D, Nolan J, Mamas MA. Radial Artery Occlusion After Transradial Interventions: A Systematic Review and Meta-Analysis. J Am Heart Assoc. 2016 Jan 25;5(1):e002686. doi: 10.1161/JAHA.115.002686. PMID 26811162
- [Result] Tehrani DM, Seto AH. Heparin, compression, and radial artery occlusion: Less is more. Catheter Cardiovasc Interv. 2021 Jun 1;97(7):1377-1378. doi: 10.1002/ccd.29764. No abstract available. PMID 34107564
- [Result] Hadjivassiliou A, Kiemeneij F, Nathan S, Klass D. Ultrasound-guided access to the distal radial artery at the anatomical snuffbox for catheter-based vascular interventions: a technical guide. EuroIntervention. 2021 Mar 19;16(16):1342-1348. doi: 10.4244/EIJ-D-19-00555. PMID 31380781
- [Result] Kiemeneij F. Left distal transradial access in the anatomical snuffbox for coronary angiography (ldTRA) and interventions (ldTRI). EuroIntervention. 2017 Sep 20;13(7):851-857. doi: 10.4244/EIJ-D-17-00079. PMID 28506941
- [Result] Soydan E, Akin M. Applicability of left distal radial artery access site in ST-segment elevation myocardial infarction; A comparative evaluation with the conventional transfemoral approach. J Vasc Access. 2022 Jan;23(1):81-87. doi: 10.1177/1129729820983138. Epub 2020 Dec 21. PMID 33349158
- [Result] Colletti G, Auslender J, De Meester A, Aminian A, Kayaert P, Ungureanu C. Feasibility and Safety of Performing Complex Coronary Interventions by Distal Radial Artery Using the Railway Sheathless Vascular System. J Invasive Cardiol. 2020 Dec;32(12):459-462. doi: 10.25270/jic/20.00201. Epub 2020 Oct 10. PMID 33035178
- [Result] Lin Y, Sun X, Chen R, Liu H, Pang X, Chen J, Dong S. Feasibility and Safety of the Distal Transradial Artery for Coronary Diagnostic or Interventional Catheterization. J Interv Cardiol. 2020 Dec 9;2020:4794838. doi: 10.1155/2020/4794838. eCollection 2020. PMID 33380922
- [Result] Tsigkas G, Papageorgiou A, Moulias A, Kalogeropoulos AP, Papageorgopoulou C, Apostolos A, Papanikolaou A, Vasilagkos G, Davlouros P. Distal or Traditional Transradial Access Site for Coronary Procedures: A Single-Center, Randomized Study. JACC Cardiovasc Interv. 2022 Jan 10;15(1):22-32. doi: 10.1016/j.jcin.2021.09.037. Epub 2021 Dec 15. PMID 34922888
- [Result] Mhanna M, Beran A, Nazir S, Al-Abdouh A, Barbarawi M, Sajdeya O, Ayesh H, Nesheiwat Z, Malhas SE, Eltahawy EA. Outcomes of distal versus conventional transradial access for coronary angiography and intervention: An updated systematic review and meta-analysis. Int J Cardiol. 2021 Dec 1;344:47-53. doi: 10.1016/j.ijcard.2021.10.003. Epub 2021 Oct 6. PMID 34626744
- [Result] Eid-Lidt G, Rivera Rodriguez A, Jimenez Castellanos J, Farjat Pasos JI, Estrada Lopez KE, Gaspar J. Distal Radial Artery Approach to Prevent Radial Artery Occlusion Trial. JACC Cardiovasc Interv. 2021 Feb 22;14(4):378-385. doi: 10.1016/j.jcin.2020.10.013. PMID 33602433
- [Result] Hamilton GW, Farouque O. Could Distal Radial Artery Access do More Than "Just" Reduce Rates of Radial Artery Occlusion? JACC Cardiovasc Interv. 2021 May 10;14(9):1042-1043. doi: 10.1016/j.jcin.2021.03.055. No abstract available. PMID 33958163
- [Derived] Li F, Zhou T, Fan X, Chen T, Shi G, Li L, Cai G. Safety and Efficacy of Distal Transradial Access in Patients With Small Diameter Distal Radial Artery: A Post Hoc Analysis of 2 Randomized Trials. Can J Cardiol. 2025 Dec 30:S0828-282X(25)01616-2. doi: 10.1016/j.cjca.2025.12.048. Online ahead of print. PMID 41478549
- [Derived] Chen T, Li L, Li F, Lu W, Shi G, Li W, Yang A, Huang H, Xiao J, Zhang Q, Gu J, Xue S, Zhang L, Li L, Xu L, Ji R, Wang H, Cai G. Comparison of long-term radial artery occlusion via distal vs. conventional transradial access (CONDITION): a randomized controlled trial. BMC Med. 2024 Feb 8;22(1):62. doi: 10.1186/s12916-024-03281-7. PMID 38331793